CLINICAL TRIAL: NCT03758326
Title: Measurement of Body Image in Eating Disorders
Brief Title: A New Measure of Body Image in Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-001-01
Record Dates: First submitted 2018-03-19; First posted 2018-11-29 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Eating Disorder
Keywords: Body image
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eating disorder (Other): Measurement of body image via Body App and relationship to body measurement
  Interventions: Other: Body App
- Healthy comparison (Other): Measurement of body image via Body App and relationship to body measurement
  Interventions: Other: Body App

INTERVENTIONS:
Other: Body App — Participants will indicate areas of concern on a virtual manikin using an electronic online interface. Body measurements will also be collected.

SUMMARY:
This study aims to compare a new electronic instrument called (here referred to as the 'Body App') with traditional paper and pencil rating scales for assessing how individuals with eating disorders evaluate their body image.

DETAILED DESCRIPTION:
Self-perceived weight or shape disturbance is a core symptom of eating disorders, with heavy therapeutic and prognostic relevance. Developing a reliable and unbiased method to assess body image disturbance is imperative, as feature characteristics of eating disorders, such as anorexia nervosa, include the overestimation of body size and shape. Among the most essential features of the disorder, this inability to correctly judge one's own body image has been frequently linked to the maintenance of eating disorders. Moreover, persistent perceptual disturbance for one's visual appearance is one of the strong predictors of relapse in AN and bulimia nervosa.

Body image disturbance can be conceptualized as having two main components: perceptual, and attitudinal/affective. These might be considered two distinct constructs, best measured independently. However, clinicians currently rely upon self-report questionnaires that evaluate aggregates of symptoms, perceptual experiences, behaviors, and thoughts linked to the disorder. Some scales selectively evaluate body image characteristics such as body dissatisfaction and body distortion. However, it is unclear to what degree each of these measures quantifies the specific components of perceptual experiences vs. attitudinal/affective aspects. This study aims to evaluate whether a new electronic instrument, here referred to as the 'Body App', which separates estimations of body shape and size from the attitudinal/affective component might result in closer approximations of the perceptual component of weight or shape disturbance, and facilitate the assessment of body image disturbance in eating disorders.

ELIGIBILITY:
Eating disorders group:

Inclusion Criteria:

* Primary clinical diagnosis of eating disorder
* Receiving inpatient treatment for eating disorder
* Body mass index greater than or equal to 14
* Independently ambulatory
* Possession of a smartphone with data plan
* English proficiency

Exclusion Criteria:

* Active suicidal ideation
* Comorbid schizophrenia spectrum or other psychotic disorder.

Healthy comparison group:

Inclusion Criteria:

* No current psychiatric diagnosis
* Body mass index greater than or equal to 14
* Independently ambulatory
* Possession of a smartphone with data plan
* English proficiency

Exclusion Criteria:

* Body mass index > 41
* Active suicidal ideation

Ages: 13 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Eligibility is based on self-representation of gender identity.
Enrollment: 135 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Body image distortion score on the Body App Tool | Through study completion, an average of 1 year
  Discrepancy between subjective body estimation on avatar and actual measurement of corresponding body part

SECONDARY OUTCOMES:
Body image dissatisfaction score on the Photographic Figure Rating Scale | Through study completion, an average of 1 year
  Average of the absolute change in body image dissatisfaction across each measurement (score range: 0 to 10; larger changes indicate greater severity of body image dissatisfaction)
Body image disturbance on the Body Appreciation Scale-2 | Through study completion, an average of 1 year
  Average of the absolute change in body image disturbance across each measurement relative to baseline (range 10 to 50, higher scores indicating reduced severity of body image disturbance)
Eating disorder severity on the Eating Disorder Examination Questionnaire | Through study completion, an average of 1 year
  Average of the absolute change in overall eating disorder severity across each measurement relative to baseline (range 0 to 6, larger scores indicate greater severity of eating disorder)
Body image disturbance on the Body Image States Scale | Through study completion, an average of 1 year
  Average of the absolute change in body image disturbance across each measurement relative to baseline (range 0 to 48, higher scores indicate greater severity of body image disturbance)
Body dysmorphic concerns on the Dysmorphic Concerns Questionnaire | Through study completion, an average of 1 year
  Average of the absolute change in dysmorphic concerns across each measurement relative to baseline (range 0 to 21, higher scores indicate greater severity of dysmorphic concerns)
Exercise addiction on the Exercise Addiction Inventory | Through study completion, an average of 1 year
  Average of the absolute change in exercise addiction across each measurement relative to baseline (range 6 to 30, higher scores indicate greater severity of exercise addiction)

CONTACTS AND LOCATIONS:
Overall Officials: Sahib Khalsa, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No